CLINICAL TRIAL: NCT02473770
Title: Rapid Acquisition of Pre and Post-Incident Disaster Data Study
Brief Title: Rapid Acquisition of Pre- and Post-Incident Disaster Data
Status: Withdrawn | Type: Observational
Why Stopped: New prepositioned protocol being developed to optimize its use in the disaster setting and broaden its reach.
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915133; 15-E-N133
Record Dates: First submitted 2015-06-13; First posted 2015-06-17 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Biological Specimens
Keywords: Registry; Exposures; Biological Specimens; Occupational Health; Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, urine, nail clippings, buccal cells, saliva, and hair.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Disaster responders: Conducting emergency disaster relief.

SUMMARY:
Background:

- Disasters like earthquakes, floods, and oil spills can give people health problems. Workers who respond to a disaster (like police and firefighters) are directly exposed to contaminants during the emergency response. So they could be at the greatest risk for these problems. Researchers want to gather data about these workers before and right after they go to a disaster. They hope this will help them understand the health effects of disasters.

Objectives:

- To answer questions about the health effects of disaster exposures. To create a participant registry and collect biological samples and health data.

Eligibility:

- People at least 21 years of age who are sent to a disaster area for an emergency response.

Design:

* Participants will have 1 study visit.
* Participants will answer questions about:
* Contact information
* Health, lifestyle, emotions
* Medical history
* Disaster response activities
* Things they are exposed to in the environment
* Participants may have blood collected from a vein in the arm.
* Participants may give biological samples. These may be urine, saliva, cheek cells, nail clippings, or hair.
* Participants will have a short physical exam. They may have their hip and waist measured over their clothes. The amount of oxygen in their blood may be measured by a sensor on a finger or ear.
* Participants may have a lung function test. They will take a deep breath and exhale strongly.
* Participants will be asked to agree to be contacted later to update contact data and learn about future studies.

DETAILED DESCRIPTION:
Disasters are frequently associated with environmental exposures and socioeconomic disruptions that may lead to short- and long-term health consequences. Disaster response workers are potentially at the greatest risk for adverse outcomes due to direct exposure to hazardous environmental contaminants during the emergency response process. The importance of conducting disaster responder research in the immediate aftermath of disasters has become widely recognized, but numerous barriers to doing so have also been recognized. The Rapid Acquisition of Pre- and Post-Incident Disaster Data (RAPIDD) protocol aims to address this gap by registering and characterizing a cohort of disaster response workers early in the disaster response phase to obtain baseline characteristics. Disaster response workers deployed to a disaster area to conduct emergency response activities will be targeted for enrollment. Disaster responders may include police, fire, and emergency medical personnel, as well as other responder groups such as public health personnel and workers involved in environmental remediation and restoration activities. The primary objective of the RAPIDD study is to create a research registry comprised of disaster response workers who are rostered before or immediately after deployment to a disaster area. Important secondary aims are to administer questionnaires and collect biological samples to characterize the cohort in a manner that will allow for future prospective analyses of associations between disaster exposures and health outcomes. In order to achieve these aims, we have developed a protocol, operational manuals, questionnaires, data collection systems, training plans, and other tools to reduce the time required to initiate disaster research. We will also obtain scientific and regulatory approval of the protocol in advance of the disaster in hopes that expedited amendments, with clarifications of the research, will minimize delays associated with various review cycles.

In order to characterize the cohort prior to their involvement with response activities that could lead to disaster-related exposures, we will attempt to collect a wide range of questionnaire data, clinical measurements and biological samples. Questionnaires may cover topics including contact information, demographics, socioeconomic status, medical history, current physical and mental health status, occupational exposures, alcohol and tobacco use and other lifestyle factors.

Biological specimens collected may include the following: blood, urine, nail clippings, saliva, buccal cells or hair. Clinical measurements may include vital signs, anthropometric measurements and spirometry. By seeking IRB and other regulatory approvals for carrying out this research in advance, we anticipate that we will be able to submit expedited amendments to clarify the research plan for a specific disaster so that research can be initiated early in the response phase. However, in the very early phases of some disaster situations, it may not be safe or feasible to collect the data needed to fully characterize a cohort of response workers. In these situations, data collection may be limited to rostering and limited self-collection of biospecimens. As the response effort stabilizes and more becomes known about potential exposures and related adverse health outcomes, we intend to expand our data collection effort, and we will seek expedited regulatory approval to do so.

ELIGIBILITY:
* INCLUSION CRITERIA:
* At least 21 years of age
* Is part of an eligible disaster responder cohort as defined in Section 5 that has received IRB approval for inclusion

EXCLUSION CRITERIA:

-Any conditions that, in the opinion of the Investigator, would pose an unacceptable risk to the participant or to the validity of the study results

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Disaster responders deployed to a disaster area to conduct emergency response activities. Disaster responders may include traditional first responders such as police, fire, and emergency medical personnel, as well as non-traditional responder groups such as public health personnel and workers involved in environmental remediation and restoration activities.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Create a research registry comprised of disaster response workers who are rostered before or immediately after deployment to a disaster area. | On going
  This is a registry study conducted to establish and characterize a cohort of disaster responders deployed to a disaster area to conductemergency response activities.

SECONDARY OUTCOMES:
Gather sociodemographic, health status, occupational exposure, and lifestyle information of the cohort before or immediately after deployment to a disaster area | Ongoing
Collect, process and store biological samples to allow estimations of disaster-related exposures of the disaster response worker cohort before or immediately after deployment to a disaster area | Ongoing
Establish a well-characterized disaster response worker cohort that will allow for future analyses of associations between disaster exposures and health outcomes | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Garantziotis, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Lurie N, Manolio T, Patterson AP, Collins F, Frieden T. Research as a part of public health emergency response. N Engl J Med. 2013 Mar 28;368(13):1251-5. doi: 10.1056/NEJMsb1209510. No abstract available. PMID 23534565